CLINICAL TRIAL: NCT06778382
Title: Deferred Systemic Therapy Following Destructive Local Treatment of Pulmonary Oligometastases After NED in Colorectal Cancer： A Phase II, Single-Arm Clinical Trail.
Brief Title: Delayed Systemic Therapy Following Destructive Local Treatment of Pulmonary Oligometastases After No Evidence of Disease (NED) in Colorectal Cancer.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinbo Yue, Director of Radiation Oncology Department, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2024-415-01
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Neoplasms Malignant
Keywords: Colorectal Neoplasms Malignant; No evidence of disease; Lung metastases; Oligometastasis; Time without systemic therapy
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oligometastasis Treatment (Experimental): including radiotherapy group, radiofrequency ablation group and surgery group
  Interventions: Combination Product: Oligometastasis Treatment

INTERVENTIONS:
Combination Product: Oligometastasis Treatment — Oligometastatic Radiotherapy Group: Patients will receive radiotherapy to lung lesions, with the lung metastases outlined as the Gross Tumor Volume (GTV). The prescribed dose will be based on a BED (Biologically Effective Dose) of 72-100 Gy, using either conventional split, macrodissected, or SBRT (Stereotactic Body Radiation Therapy) at the investigator's discretion. No systemic therapy will be administered.
  Oligometastatic Radiofrequency Ablation Group: For lesions suitable for radiofrequency ablation, this will be performed in consultation with the Department of Interventional Medicine, considering patient and family preferences. Systemic therapy will not be given.
  Oligometastatic Surgery Group: For lesions suitable for surgical resection, patients will undergo surgery after consultation with the Department of Surgery. No systemic therapy will be performed.

SUMMARY:
Colorectal cancer (CRC) is the third most common cancer worldwide. Surgical resection is one of the primary treatment options for CRC; however, postoperative recurrence remains a significant clinical challenge for both the medical community and patients. Postoperative chemotherapy, as an important adjuvant therapy, is widely used in CRC patients aiming to reduce the risk of recurrence. Despite extensive research on the efficacy of postoperative chemotherapy in CRC, the mechanisms of postoperative recurrence, predictive factors, and strategies to enhance chemotherapy effectiveness remain unclear. For colorectal cancer patients who have achieved NED (No Evidence of Disease), the decision to either reinitiate or change the systemic chemotherapy regimen for newly developed pulmonary oligometastases remains controversial. Local treatment options for diagnosing oligometastases include surgery, radiotherapy, and radiofrequency ablation. However, whether systemic treatment should be added after local treatment in patients who have achieved NED remains uncertain , and this issue requires urgent resolution.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common cancer worldwide. Surgical resection is a primary treatment option; however, postoperative recurrence remains a significant challenge. Postoperative chemotherapy is commonly used as an adjuvant treatment to reduce recurrence risk, but the mechanisms of recurrence, predictive factors, and strategies to enhance chemotherapy efficacy remain unclear.For CRC patients who have achieved No Evidence of Disease (NED), the decision to reinitiate or modify systemic chemotherapy for newly developed pulmonary oligometastases is still debated. Local treatment options for pulmonary oligometastases include surgery, radiotherapy, and radiofrequency ablation. However, whether systemic therapy should follow local treatment in NED patients is uncertain.This issue is actively debated in multidisciplinary team (MDT) consultations both in our hospital and across the country. Some experts argue that pulmonary oligometastases signify disease progression, requiring systemic treatment, while others suggest that these metastases may not indicate high malignancy and that observation, with possible delayed systemic treatment, could be sufficient.This study will include CRC patients who have achieved NED for at least six months and then develop pulmonary oligometastases, treated exclusively with destructive local therapies (surgery, radiotherapy, or ablation) without systemic therapy. The study will assess the timing of transitioning to the next line of systemic therapy through imaging and ctDNA monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a pathologically confirmed diagnosis of colorectal cancer with the following disease conditions:

  1. The patient has achieved No Evidence of Disease (NED) after undergoing EMR, surgery, radiofrequency ablation, or radiotherapy.
  2. NED has been maintained for ≥ 6 months.
  3. The patient has not received chemotherapy, or has only received postoperative adjuvant chemotherapy or first-line systemic therapy.
  4. Oligometastatic lung lesions (defined as 5 or fewer lesions) detected after ≥ 6 months of NED maintenance, eligible for destructive therapy.
  5. No prior radiotherapy to the lungs.
* RECIST 1.1 criteria: The patient must have measurable lesions, defined as at least one nodal lesion with a longest diameter > 1.5 cm, or at least one nodal lesion > 1 cm with an accurately measurable pendulous diameter.
* ECOG performance status: ≤ 2 (Eastern Cooperative Oncology Group general condition score).
* The patient's expected survival must be ≥ 3 months.
* Adequate hematologic function: Absolute neutrophil count ≥ 1.6 x 10⁹/L, with no growth factor support for at least 7 days prior to testing.
* Normal organ function: The patient must be able to tolerate at least one of the local destructive treatments, as assessed by the corresponding department's physician, based on normal hepatic, renal, pulmonary, and cardiac function.
* Reproductive age: Female patients of childbearing potential must agree to use a reliable method of contraception with their partner from the time of informed consent until 1 year after treatment completion.
* The patient must have voluntarily provided informed consent to participate in the study.

Exclusion Criteria:

* First diagnosis of advanced colorectal cancer with metastatic disease.
* Multiple lung metastases (> 5 lesions), liver metastasis, bone metastasis, or lymph node metastasis.
* Lung metastases that are not amenable to radiotherapy, as determined by the investigator.
* Previously received second-line or higher systemic treatment.
* Liver or kidney dysfunction: Alanine aminotransferase (ALT) > 3 times the upper limit of normal; Aspartate aminotransferase (AST) > 3 times the upper limit of normal; Total bilirubin (TBIL) > 2 times the upper limit of normal; Serum creatinine > 1.5 times the upper limit of normal.
* Elevated tumor marker: CEA ≥ 50 ng/mL.
* Serious medical conditions that may interfere with the study (e.g., uncontrolled diabetes, gastric ulcers, severe cardiopulmonary diseases), at the discretion of the researchers.
* Severe or uncontrolled infections.
* Active autoimmune disease.
* Clinically significant central nervous system dysfunction.
* Recent major surgery (excluding lymph node biopsy) within the last 30 days.
* Pregnant or breastfeeding women of childbearing age who are not using contraception.
* Drug allergy to study treatments.
* Other reasons, as determined by the researchers, that make the patient unsuitable for participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Time Without Systemic Therapy | 2 years
  The time interval between diagnosis or the completion of the current systemic treatment and the start of the next systemic therapy

SECONDARY OUTCOMES:
Progression-Free Survival（PFS） | 2 years
  The time interval between enrollment and disease progression or death for patients in the intent-to-treat population, whichever occurred first. For those who did not progress at the time of withdrawal from the trial or whose time to disease progression was not recorded, the date of the last examination was used as the endpoint date
Time to Next Treatment (TTNT) | 2 years
  The time interval from the completion of the first SBRT/radiofrequency ablation/surgery to the initiation of the next anticancer treatment or death from any cause
Overall Response Rate (ORR) | 2 years
  Percentage of subjects in the protocol-eligible population and in the intent-to-treat population who achieved CR+PR after treatment
Disease Control Rate (DCR) | 2 years
  Percentage of subjects in the protocol-eligible population and in the intention-to-treat population who achieved CR+PR+SD after treatment
Complete Response Rate (CRR) | 2 years
  Percentage of subjects achieving CR after treatment in the protocol-eligible population as well as in the intent-to-treat population
Duration of Response (DOR) | 2 years
  The time from the start of the first assessment of the tumor as CR or PR to the first assessment of PD or death from any cause
Overall Survival (OS) | 2 years
  The time interval between enrollment and death for patients in the intent-to-treat (ITT) population. If the patient continues to be alive or his/her fate is unknown, the date of death will be the most recent point in time at which the patient was known to be alive
Incidence of Adverse Effects | 2 years
  Evaluation of toxicity according to NCI CTCAE 5.0 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jinbo Yue, Dorcter, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Department of Radiation Oncology, Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horie T, Kanemitsu Y, Takamizawa Y, Moritani K, Tsukamoto S, Shida D. Prognostic differences between oligometastatic and polymetastatic disease after resection in patients with colorectal cancer and hepatic or lung metastases: Retrospective analysis of a large cohort at a single institution. Surgery. 2023 Feb;173(2):328-334. doi: 10.1016/j.surg.2022.10.014. Epub 2022 Nov 15. PMID 36400583
- [Background] Benson AB, Venook AP, Adam M, Chang G, Chen YJ, Ciombor KK, Cohen SA, Cooper HS, Deming D, Garrido-Laguna I, Grem JL, Haste P, Hecht JR, Hoffe S, Hunt S, Hussan H, Johung KL, Joseph N, Kirilcuk N, Krishnamurthi S, Malla M, Maratt JK, Messersmith WA, Meyerhardt J, Miller ED, Mulcahy MF, Nurkin S, Overman MJ, Parikh A, Patel H, Pedersen K, Saltz L, Schneider C, Shibata D, Shogan B, Skibber JM, Sofocleous CT, Tavakkoli A, Willett CG, Wu C, Gurski LA, Snedeker J, Jones F. Colon Cancer, Version 3.2024, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2024 Jun;22(2 D):e240029. doi: 10.6004/jnccn.2024.0029. PMID 38862008
- [Background] Loft M, To YH, Gibbs P, Tie J. Clinical application of circulating tumour DNA in colorectal cancer. Lancet Gastroenterol Hepatol. 2023 Sep;8(9):837-852. doi: 10.1016/S2468-1253(23)00146-2. Epub 2023 Jul 24. PMID 37499673
- [Background] Wang K, Wang X, Pan Q, Zhao B. Liquid biopsy techniques and pancreatic cancer: diagnosis, monitoring, and evaluation. Mol Cancer. 2023 Oct 6;22(1):167. doi: 10.1186/s12943-023-01870-3. PMID 37803304
- [Background] Abbosh C, Hodgson D, Doherty GJ, Gale D, Black JRM, Horn L, Reis-Filho JS, Swanton C. Implementing circulating tumor DNA as a prognostic biomarker in resectable non-small cell lung cancer. Trends Cancer. 2024 Jul;10(7):643-654. doi: 10.1016/j.trecan.2024.04.004. Epub 2024 Jun 4. PMID 38839544
- [Background] Tao XY, Li QQ, Zeng Y. Clinical application of liquid biopsy in colorectal cancer: detection, prediction, and treatment monitoring. Mol Cancer. 2024 Jul 16;23(1):145. doi: 10.1186/s12943-024-02063-2. PMID 39014366
- [Background] Gouda MA, Janku F, Wahida A, Buschhorn L, Schneeweiss A, Abdel Karim N, De Miguel Perez D, Del Re M, Russo A, Curigliano G, Rolfo C, Subbiah V. Liquid Biopsy Response Evaluation Criteria in Solid Tumors (LB-RECIST). Ann Oncol. 2024 Mar;35(3):267-275. doi: 10.1016/j.annonc.2023.12.007. Epub 2023 Dec 23. PMID 38145866